CLINICAL TRIAL: NCT01968759
Title: A Prospective, Randomized, Multicenter, Open, Blinded Endpoint (PROBE), Clinical Trial to Assess the Renal and Humoral Effects of Sevelamer Carbonate in Patients With Chronic Kidney Disease and Residual Proteinuria Despite Best Available Treatment
Brief Title: Sevelamer in Proteinuric CKD
Acronym: ANSWER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANSWER; 2012-005416-26 (EudraCT Number)
Record Dates: First submitted 2013-10-15; First posted 2013-10-24 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Sevelamer carbonate; Proteinuria; Phosphate binders
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Sevelamer; Ramipril; Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramipril and Irbesartan (Active Comparator): Best available therapy including dual RAS blockade with Ramipril and Irbesartan
  Interventions: Drug: Sevelamer; Drug: Ramipril and Irbesartan
- Sevelamer (Experimental): Two tablets of Sevelamer carbonate 800 mg will be orally administered three times per day during the meals for 3 months.
  Interventions: Drug: Sevelamer; Drug: Ramipril and Irbesartan

INTERVENTIONS:
Drug: Sevelamer
Drug: Ramipril and Irbesartan

SUMMARY:
Progressive renal impairment in chronic kidney diseases (CKD) may cause inability to excrete phosphate load, thus leading to the typical abnormalities of the mineral metabolism, such as increased phosphate and reduced calcium levels, 1,25- dihydroxyvitamin D deficiency and secondary hyperparathyroidism (HPT). Treatment with vitamin D analogues and/or phosphate binders ameliorates these abnormalities that are also associated with accelerated renal disease progression and increased cardiovascular risk. However in a post-hoc analysis of 331 patients with proteinuric chronic nephropathies included in the Ramipril Efficacy In Nephropathy (REIN) trial, increasing serum phosphate levels at inclusion, even within the normal reference range, were associated with an incremental risk of progression to End Stage Renal Disease (ESRD). Moreover, increasing levels of serum phosphate were associated with a progressively decreasing protective effect of ramipril therapy against progression to ESRD, to the point that the benefit of Angiotensin-Converting-Enzyme (ACE) inhibition was almost fully lost among patients with serum phosphate levels exceeding 4.5 mg/dL. This finding provided convincing evidence that phosphate plays a direct pathogenic role in patients with progressive nephropathies and that excess phosphate exposure may limit or even blunt the renoprotective effect of ACE inhibitor therapy in this population.

Sevelamer carbonate is a newly approved phosphate binder for chronic kidney disease (CKD) patients not yet on maintenance dialysis. Treatment with Sevelamer, in addition to correct hyperphosphatemia, was also found to ameliorate abnormalities of the mineral metabolism associated with accelerated renal disease progression and increased cardiovascular risk. Moreover, Sevelamer therapy reduces proteinuria in an animal model of uremia, an effect that in the long term might translate into significant renoprotection. These findings suggest that serum phosphate might be a specific target for renoprotective therapy in CKD patients and provide the background for randomized clinical trials to formally test whether reducing phosphate exposure by phosphate binding agents may serve to optimize the renoprotective effect of RAS inhibition in this population. Thus, whether phosphate reduction by Sevelamer carbonate therapy may have a specific antiproteinuric effect in humans with chronic nephropathies and residual proteinuria despite optimized RAS inhibitor therapy is worth investigating.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* estimated glomerular filtration rate (GFR) by simplified MDRD formula > 15 mL/min/1.73m2;
* 24-h urinary protein excretion rate ≥ 0.5 g/24hour;
* no concomitant treatment with phosphate binders;
* written informed consent

Exclusion Criteria:

* serum phosphate level < 2.5 or > 5.5 mg/dL;
* patients with serum PTH levels >250 pg/mL without stable vitamin D (calcitriol or paricalcitol) or calcimimetics therapy from at least three months;
* serum calcium level < 7.5 or >10.5 mg/dL;
* history of congestive heart failure, myocardial infarction, cerebrovascular accident within the last 6 months;
* cancer and any severe systemic disease or clinical condition that may jeopardize data interpretation or completion of the study;
* presence of, or predisposition to, intestinal or ileus obstruction or severe gastrointestinal motility disorder (like severe constipation);
* previous major gastrointestinal surgery;
* previous kidney transplantation;
* previous parathyroidectomy;
* concomitant treatment with antiacid and phosphate binders with aluminium, magnesium, calcium or lanthanum;
* pregnancy or breastfeeding;
* childbearing potential without reliable contraceptive methods during the whole study period;
* participation in any clinical trial using an investigational product or device during the 30 days preceding the first protocol visit;
* alcohol or drug (excluding tobacco) abuse ;
* inability to comply with the study procedures during the whole study period, legal incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
24-h urinary protein excretion | Changes from Baseline at 3,4,7 and 8 month.

SECONDARY OUTCOMES:
Office blood pressure | At every visit, up to 8 months.
Glomerular Filtration Rate | Changes from baseline at 3,4 and 7 month.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Clinical Research Center for Rare Diseases, Ranica, Bergamo
  - Azienda Ospedaliera "Bianchi-Melacrino-Morelli" c/o Ospedali Riuniti U.O. Nefrologia, Dialisi e Trapianto, Reggio Calabria, Reggio Calabria

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Ruggiero B, Trillini M, Tartaglione L, Rotondi S, Perticucci E, Tripepi R, Aparicio C, Lecchi V, Perna A, Peraro F, Villa D, Ferrari S, Cannata A, Mazzaferro S, Mallamaci F, Zoccali C, Bellasi A, Cozzolino M, Remuzzi G, Ruggenenti P, Kohan DE; ANSWER Study Organization. Effects of Sevelamer Carbonate in Patients With CKD and Proteinuria: The ANSWER Randomized Trial. Am J Kidney Dis. 2019 Sep;74(3):338-350. doi: 10.1053/j.ajkd.2019.01.029. Epub 2019 Apr 23. PMID 31027883